CLINICAL TRIAL: NCT05109468
Title: Assessment of Patients' Quality of Sexual Life After Anal Cancer Treatment
Acronym: SEQUOIA
Status: Active, not recruiting | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PROICM 2021-03 OSE
Record Dates: First submitted 2021-10-04; First posted 2021-11-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Anal Cancer; Sexuality; Psychologic Stress; HPV; Anxiety
MeSH Terms: conditions — Anus Neoplasms; Sexuality; Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anal cancer patients: Non-metastatic squamous anus cancer with the presence of an HPV infection authenticated on the biopsy
  Interventions: Other: Quality of life questionnaire

INTERVENTIONS:
Other: Quality of life questionnaire — to assess the quality of sexual life of patients treated for anal cancer treated with radiotherapy, during their treatment, then 3 months after treatment and, finally, 2 years after cancer diagnosis.

SUMMARY:
The purpose of this this study, to evaluate the quality of sexual life of patients treated for anal cancer treated by radiotherapy, during their treatment, then 3 months after treatment and, finally, 2 years after treatment. cancer diagnosis.

DETAILED DESCRIPTION:
Sexual health is defined by WHO in 2011 as a state of physical, emotional, mental and social well-being in relation to sexuality. It is an integral part of health, well-being and quality of life and is recognized as a right of everyone.Alteration of sexuality after cancer impacts all phases of the sexual response. It is multifactorial: psychological (ie, anxiety linked to the disease, fear of death, or impairment of body image) and physiological (ie, alteration of the sexual reaction which may be linked, in part, to direct sequelae generated by irradiation of the genitals).

Anal cancer remains fairly rare, affecting around 2,200 people each year in France, with a predominance of women (60 to 70% of patients), However, its incidence has been growing strongly for 30 years, in Europe and the United States where it is has increased by 70% over the last 10 years alone, in both men and women, with an increasingly younger population.

It is linked, in more than 90% of cases, to a carcinogenic virus, the Human PapillomaVirus (HPV), a late consequence of an infection, most often asymptomatic, transmitted by the sexual route.

The question of sexuality after cancer remains, in fact, very little addressed by doctors who express a lack of training. Patients, for their part, often do not dare to raise the issue with caregivers, out of modesty, or thinking that the teams do not have the time. Discussions with patients therefore generally always remain focused on oncological management, from the initial consultation to the follow-up consultations. The hope of recovery awaited on each of the assessments and the fear of relapse often obscure more global and equally essential questions: whether it is about the quality of life, the after-effects, or even more, the quality. of sex life. For these reasons, this study will collect the information provided to patients on the impact of this treatment on their sexual health, whether it is medical information recorded in the file, or information perceived and retained by patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years old.
2. Patient treated for non-metastatic squamous cell anus cancer with the presence of an HPV infection authenticated on the biopsy.
3. Patient living with a partner or having an active sex life the year preceding the diagnosis.
4. Patient who, after information, agrees to participate in the study.
5. Patient affiliated to a French social security scheme.

Exclusion Criteria:

1. Patient unable or unwilling to complete a questionnaire on the quality of sexual life.
2. Patient without sexual activity the year before diagnosis.
3. Patient whose regular follow-up is impossible for psychological, family, social or geographic reasons.
4. Patient under guardianship, curatorship or legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This project is a descriptive study without formal calculation of the number of subjects required. The sample size will be based on the ability to recruit at the ICM over a 30-month period.
  The active queue of patients at the ICM is about 3 to 4 patients per month, with an estimate of the proportion of refusals expected at 50% in these patients still on the shock of the announcement of cancer, where the theme of sexuality does not always appear essential at this time.
  Recruiting 50 patients would make it possible to have an estimate (for descriptive purposes) of the mean scores after treatment (visit 3 months after treatment) on the EORTC SHQ-C22 quality of sexual life questionnaire (the range of which goes from 0 to 100 ), with a level of precision of 12.25 (amplitude of the confidence interval) for a two-sided 95% confidence interval and a standard deviation of 22.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Change in Sexual quality of life score | at inclusion, 3 months post-treatment and 2 years after the announcement of cancer.
  Sexual quality of life score obtained on the European EORTC SHQ-C22 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claire LEMANSKI, MD, Study Chair — Institut Régional du Cancer de Montpellier
Locations (1):
- Institut régional du Cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No